CLINICAL TRIAL: NCT03680911
Title: Early N-Acetyl Cysteine Treatment for Head Trauma-induced Anosmia
Brief Title: NAC for Head Trauma-induced Anosmia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor participant compliance
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Roy R. Casiano, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170856
Record Dates: First submitted 2018-08-29; First posted 2018-09-21 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Anosmia; Head Trauma
MeSH Terms: conditions — Anosmia; Craniocerebral Trauma | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC Group (Experimental): NAC group will be administered orally as a 4 gram loading dose, followed by 2 g PO BID for 4 days, then 1.5 g PO BID for 2 days
  Interventions: Drug: N Acetyl Cysteine
- Placebo Group (Placebo Comparator): Placebo group will be administered orally as a 4 gram loading dose, followed by 2 g PO BID for 4 days, then 1.5 g PO BID for 2 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: N Acetyl Cysteine — 2 g PO BID for 4 days, then 1.5 g PO BID for 2 days
  Arms: NAC Group
Drug: Placebo oral capsule — 2 g PO BID for 4 days, then 1.5 g PO BID for 2 days
  Arms: Placebo Group

SUMMARY:
This study will compare administration of N-Acetyl Cysteine (NAC) versus placebo for the treatment of olfactory loss due to head injury. The hypothesis is that treatment with NAC acutely after head injury will result in improved olfactory function

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Ryder Trauma Center for observation acutely following head injury (i.e. concussion), with documented hyposmia or anosmia by University of Pennsylvania Smell Identification Test (SIT).
* Male or female, aged 18 years or older
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Ability to take oral medication and be willing to adhere to the NAC regimen
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of NAC administration

Exclusion Criteria:

* Severe trauma requiring ongoing inpatient treatment beyond 48 hours
* Pregnancy (based on urine screening) or lactation
* Known allergic reactions to components of NAC, such as Mucomyst
* Currently taking nitrates such as nitroglycerine and/or isosorbide regularly
* Currently taking azathioprine (Imuran) or cyclophosphamide (Cytoxan)
* Known diagnosis of cystinuria (renal condition in which cysteine supplement should be avoided)
* Febrile illness within 1 week
* Treatment with another investigational drug or other intervention within 3 months
* Active sinonasal disease by imaging and/or nasal exam, i.e. rhinosinusitis, nasal polyps
* Adults unable to consent
* Prisoners, employees or subordinates
* Individuals who are not yet adults (infants, children, teenagers). This population is excluded because efficacy has not yet been established in adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Casiano, MD, Principal Investigator — University of Miami
Locations (1):
- University Of Miami, Otolaryngology Department, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Visit 1 (Baseline)
Arm/Group | NAC Group | Placebo Group
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: At Home Treatment
Arm/Group | NAC Group | Placebo Group
Started | 3 | 4
Completed | 0 | 1
Not Completed | 3 | 3
Not completed — Study Termination | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Visit 2 (1 Month Follow up)
Arm/Group | NAC Group | Placebo Group
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: Visit 3 (4 Month Follow up)
Arm/Group | NAC Group | Placebo Group
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Study Termination | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAC Group | Placebo Group | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.9) | 36.8 (15.8) | 41.7 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Olfactory Function
Description: Olfactory function will be measured using the University of Pennsylvania Smell Identification Test (UPSIT). The UPSIT is a self-administered 40-item test involving microencapsulated (scratch-and-sniff) odors with a forced-choice design. The total score ranges from 0-40 with the higher score indicating better olfactory function.
Time Frame: 4 months
Population: Data will not be reported due to confidentiality, there was only one participant to complete the 1 month follow up visit. Study was terminated prior to the remaining participants completing any follow up visits as per protocol.
Arm/Group | NAC Group | Placebo Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life Questionnaire
Description: Quality of life will be measured using the questionnaire for Olfactory Disorders (QOD). QOD has a total score from 0-75 with the higher score indicating a better quality of life.
Time Frame: 4 months
Population: as for outcome 1
Arm/Group | NAC Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 weeks
Description: Only treatment-related adverse events are collected and reported. Non-treatment related Adverse Events were not monitored/assessed.
Arm/Group | NAC Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03680911/Prot_SAP_000.pdf